CLINICAL TRIAL: NCT01314768
Title: RCT of Structured Brief Intervention for Medication Overuse Headache Versus Business as Usual
Brief Title: Brief Intervention for Medication Overuse Headache
Acronym: BIMOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Christofer Lundqvist, Principal investigator/Project leader, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIMOH
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Medication-overuse Headache; Chronic Headache
MeSH Terms: conditions — Headache Disorders, Secondary; Headache Disorders | interventions — Crisis Intervention; Commerce; Mass Screening

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Brief intervention (Active Comparator): Behavioural brief intervention delivered by GP
  Interventions: Behavioral: Brief intervention
- Business as usual (Placebo Comparator): Business as usual according to individual GP
  Interventions: Other: Business as usual
- Chronic headache control (Other): Screening and outcome control only. Non-intervention Control, screened and followed-up at final time point
  Interventions: Other: Screening and outcome evaluation only
- Population control (Other): Screening and outcome control only. Non-intervention Control, screened and followed-up at final time point
  Interventions: Other: Screening and outcome evaluation only

INTERVENTIONS:
Behavioral: Brief intervention — Structured behavioural Brief intervention given by trained GPs
  Arms: Brief intervention
Other: Business as usual — GPs to treat patient as they have until now based on best established practice
  Arms: Business as usual
Other: Screening and outcome evaluation only — No additional intervention
  Arms: Chronic headache control
Other: Screening and outcome evaluation only — No additional intervention
  Arms: Population control

SUMMARY:
The investigators will perform a cluster randomised controlled study of Brief intervention (BI) for medication-overuse headache (MOH) versus business as usual. GPs will be trained to perform a structured brief intervention after identifying patients with probable MOH using the severity of dependence scale. The control arm will include patients of GPs who have not been trained in BI. Patients will be recruited by prior short postal screening of patients listed on the GPs patient lists.

The hypothesis is that BI will lead to improvement of medication-overuse and chronic headache as compared to no BI.

Main outcomes are:

* number of medication days per month
* number of headache days per month
* headache index

DETAILED DESCRIPTION:
123 cases in all included (75 in intervention/placebo control arms and 48 in non-intervention Control arms) 19 did not meet predefined inclusion criteria for the different arms (5 and 8 in intervention arm and placebo arm respectively, 4 and 2 in chronic headache Control and population Control respectively)

1 case was lost to follow up in each of the 4 Groups prior to first assessment. Thus 60 cases remained in intervention/placebo Control arms (24 in intervention and 36 in placebo Control) and 40 in non intervention Control arms (15 chronic headache Controls, 25 population Controls).

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Screening positive for possible chronic headache (> 10 headache days per month) (not for population control arm)
* Screening positive for possible medication-overuse (> 15 medication days per month) (not for chronic headache control arm)

Exclusion Criteria:

* Other complicating pain with medication treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of medication days per month | 3 months
Number of headache days per month | 3 months

SECONDARY OUTCOMES:
Proportion significantly improved | 3 month
  proportion improved >50% and >25% in terms of no headache days/month
Headache medication days per month (diary reported) | 3 months
Headache days/month (diary reported) | 3 months
Average headache intensity (VAS) | 3 months
Quality of life | 3 months
Self-reported health related costs | 3 months
Long term follow up of same outcomes as above plus relapse rate | 12 months
Headache index | 3 months
  Headache intensity x frequency x duration
Follow up of same outcomes as for 3 months | 6 months
  Added extra time point due to cross over of non-treated patients into intervention Group if intervention was positive at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christofer Lundqvist, MD, PhD, Principal Investigator — Akershus University Hospital and University of Oslo
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Dept of general medicine, University of Oslo, Oslo

REFERENCES:
- [Derived] Lundqvist C, Gossop M, Russell MB, Straand J, Kristoffersen ES. Severity of Analgesic Dependence and Medication-overuse Headache. J Addict Med. 2019 Sep/Oct;13(5):346-353. doi: 10.1097/ADM.0000000000000504. PMID 30724760
- [Derived] Kristoffersen ES, Straand J, Benth JS, Russell MB, Lundqvist C. Predictors of successful primary care detoxification treatment for medication-overuse headache. Acta Neurol Scand. 2017 Nov;136(5):486-494. doi: 10.1111/ane.12759. Epub 2017 Mar 28. PMID 28369734
- [Derived] Kristoffersen ES, Straand J, Vetvik KG, Benth JS, Russell MB, Lundqvist C. Brief intervention by general practitioners for medication-overuse headache, follow-up after 6 months: a pragmatic cluster-randomised controlled trial. J Neurol. 2016 Feb;263(2):344-353. doi: 10.1007/s00415-015-7975-1. Epub 2015 Dec 8. PMID 26645391
- [Derived] Kristoffersen ES, Straand J, Russell MB, Lundqvist C. Disability, anxiety and depression in patients with medication-overuse headache in primary care - the BIMOH study. Eur J Neurol. 2016 Jan;23 Suppl 1:28-35. doi: 10.1111/ene.12850. PMID 26563095
- [Derived] Kristoffersen ES, Straand J, Vetvik KG, Benth JS, Russell MB, Lundqvist C. Brief intervention for medication-overuse headache in primary care. The BIMOH study: a double-blind pragmatic cluster randomised parallel controlled trial. J Neurol Neurosurg Psychiatry. 2015 May;86(5):505-12. doi: 10.1136/jnnp-2014-308548. Epub 2014 Aug 11. PMID 25112307
- [Derived] Kristoffersen ES, Straand J, Benth JS, Russell MB, Lundqvist C. Study protocol: brief intervention for medication overuse headache--a double-blinded cluster randomised parallel controlled trial in primary care. BMC Neurol. 2012 Aug 10;12:70. doi: 10.1186/1471-2377-12-70. PMID 22883540